CLINICAL TRIAL: NCT00719368
Title: Quantitative Sensory Testing in Persistent Postherniotomy Pain Patients
Brief Title: Neurophysiological Characterization of Postherniotomy Pain
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, M.D., Rigshospitalet, Denmark
Other Study IDs: KF 01267755
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2012-10

CONDITIONS: Postoperative Pain; Postherniotomy Pain; Neuropathic Pain
Keywords: Groin hernia; pain; chronic; quantitative sensory testing; Persistent postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Neuralgia; Hernia, Inguinal; Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pain-free control: Pain-free controls from previous prospective study (KF 01294867), operated >2 years previously
- Pain Patients: Patients with persistent postherniotomy pain lasting >1 year and pain related impaired daily function

SUMMARY:
Sensory function is different in persistent postherniotomy pain patients than in operated controls, suggesting this to be a neuropathic pain syndrome. By performing quantitative sensory testing, the specific changes in pain patients will be revealed, thereby aiding in designing future treatment trials. MRI scans of the groin regions in pain patients and control patients will be evaluated by senior MRI specialists assessing potential pathology to the region (Mesh, inflammation, edema, funicle etc.) Assessors will be blinded to clinical status, and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male patients >18 yrs
* Inguinal herniotomy >1 yr previously
* No sign of hernia recurrence
* Unilateral chronic groin pain lasting more than 3 months
* Moderate/severe pain related impairment of everyday activities.

Exclusion Criteria:

* Other causes of persistent pain in groin region (hip, other surgical procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: persistent posthenriotomy patients
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Sensory function | actual

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, M.D., Study Director — Rigshospitalet, Copenhagen University, Denmark; Henrik Kehlet, M.D., Ph. D., Principal Investigator — Rigshospitalet, Copenhagen University, Denmark
Locations (2):
- Denmark (2):
  - Danish Pain Research Centre, Aarhus
  - Section for Surgical Pathophysiology, Copenhagen

REFERENCES:
- [Background] Aasvang EK, Brandsborg B, Christensen B, Jensen TS, Kehlet H. Neurophysiological characterization of postherniotomy pain. Pain. 2008 Jul;137(1):173-181. doi: 10.1016/j.pain.2007.09.026. Epub 2007 Oct 31. PMID 17976914
- [Background] Aasvang E, Kehlet H. Chronic postoperative pain: the case of inguinal herniorrhaphy. Br J Anaesth. 2005 Jul;95(1):69-76. doi: 10.1093/bja/aei019. Epub 2004 Nov 5. No abstract available. PMID 15531621